CLINICAL TRIAL: NCT00937235
Title: Treatment of Smoking Among Individuals With PTSD: A Phase II, Randomized Study of Varenicline and Cognitive Behavioral Therapy
Brief Title: Treatment of Smoking Among Individuals With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA023507 (NIH); R01DA023507 (NIH)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Cigarette Smoking; Nicotine Dependence; Post-traumatic Stress Disorder; Tobacco Use Disorder
Keywords: Smoking Cessation; Anxiety; Behavior Therapy; Varenicline
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Stress Disorders, Post-Traumatic; Smoking Cessation; Anxiety Disorders | interventions — Varenicline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Treatment (Experimental): Prolonged Exposure + Varenicline + Medication Management Counseling
  Interventions: Drug: Varenicline; Behavioral: Medication Management Counseling; Behavioral: Prolonged Exposure
- Varenicline (Active Comparator): Varenicline + Medication Management Counseling
  Interventions: Drug: Varenicline; Behavioral: Medication Management Counseling

INTERVENTIONS:
Drug: Varenicline — 1 mg tablets, orally, twice daily x 12 weeks
  Other Names: Chantix
Behavioral: Medication Management Counseling — 15-minutes weekly counseling x 12 weeks, focused on medication adherence and smoking cessation
Behavioral: Prolonged Exposure — 75-90 minute weekly psychotherapy sessions x 12 weeks, focused on gradually confronting distressing trauma-related memories and reminders
  Other Names: Cognitive-Behavioral Therapy
  Arms: Integrated Treatment

SUMMARY:
This study will examine the effect of combining prolonged exposure, a cognitive-behavioral treatment program for post-traumatic stress disorder (PTSD) with medication (varenicline) and counseling treatments for smoking cessation. Subjects will be randomly assigned to a 3-month treatment of either: 1) varenicline and smoking cessation counseling alone, or 2) prolonged exposure, varenicline, and smoking cessation counseling. Assessments will be completed at the end of treatment and 6-month follow-up.

We hypothesize that, at the end of treatment and at follow-up, abstinence rates and decrease in cigarettes smoked will be greater among participants who receive the combined treatment for both PTSD and smoking.

ELIGIBILITY:
Inclusion Criteria:

* Male or female treatment-seeking cigarette smokers between 18-75 years old who smoke an average of ≥10 cigarettes/day during past year;
* Current diagnosis of chronic PTSD (symptom duration > 3 months) with clinically significant trauma-related symptoms (PSS-I >= 20)
* Live a commutable distance to the University of Pennsylvania and agree to follow-up visits;
* Agree not to use other forms of smoking cessation treatment or treatment for PTSD during the study period;
* If taking SRIs or other medications at intake, have been on stable medication and dose regimen for past 3 months and agree to maintain current regimen if possible;
* Demonstrate the capacity to provide informed consent;
* Speak and read English.

Exclusion Criteria:

* History of drug or alcohol abuse or dependence in past 3 months or any unwillingness to not smoke marijuana during the first 13 weeks of the study;
* Current and continuing intimate relationship with a physically or sexually abusive partner;
* Current suicidal ideation with intent and/or plan that, in the judgment of the investigator, should be the focus of treatment;
* Prior serious suicide attempt, as judged by the evaluator to have a high degree of lethality;
* Current or past history of psychosis (bipolar disorder or schizophrenia);
* History of significant cardiovascular disease or uncontrolled hypertension in past 6 months;
* Women who are pregnant, likely to become pregnant (i.e., sexually active and not using contraception), or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edna B Foa, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Dept of Psychiatry, Center for Treatment and Study of Anxiety, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center for the Treatment and Study of Anxiety — http://www.med.upenn.edu/ctsa/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements and referrals to the University of Pennsylvania's Center for the Treatment and Study of Anxiety (CTSA), Transdisciplinary Tobacco Use Research Center (TTURC), and the Philadelphia VA Hospital.
Period: Overall Study
Arm/Group | Integrated Treatment | Varenicline
Started | 72 | 70
Completed | 72 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Treatment | Varenicline | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 70 | 142
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.7) | 42.6 (10.2) | 42.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 46 | 40 | 86
Region of Enrollment [Number; unit: participants]
  United States | 72 | 70 | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point Prevalence Smoking Abstinence
Description: Number of participants reporting seven-day point prevalence abstinence (PPA), which was defined as self-reported abstinence for 7 days prior to the assessment, serum cotinine level of <15ng/ml, and CO < 10 ppm.
Time Frame: At 3-month follow-up (6-month post-quit day)
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Participants | 8 | 11

2. Secondary Outcome: Blood Serum Cotinine
Description: Level of cotinine in blood
Time Frame: At end of 3-month follow-up
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
ng/mL | 156.0 (119.4) | 149.2 (149.6)

3. Secondary Outcome: Posttraumatic Symptom Scale Interview (PSS-I) at Post-Treatment
Description: Posttraumatic Symptom Scale Interview at post-treatment assessment, which measures severity of post-traumatic stress disorder (PTSD) symptoms Total scores are displayed and represent summed scores on 17 individual items the scale, and scale range for total scores is 0 to 51.
  Higher scores indicate higher/worse levels of PTSD.
Time Frame: Post-treatment, occurring 12 weeks after the start of treatment (week 0)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Scores on a scale | 11.19 (10.63) | 18.84 (11.59)

4. Secondary Outcome: Posttraumatic Symptom Scale Interview (PSS-I) Total Score at 3-Month Follow-Up
Description: Posttraumatic Symptom Scale Interview at 3-month follow-up assessment, which measures severity of post-traumatic stress disorder (PTSD) symptoms Total scores are displayed and represent summed scores on 17 individual items the scale, and scale range for total scores is 0 to 51.
  Higher scores indicate higher/worse levels of PTSD.
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
scores on a scale | 10.35 (11.73) | 16.74 (12.11)

5. Secondary Outcome: Hamilton Depression Scale (HAM-D) Total Score at Post-Treatment
Description: Hamilton Depression scale (HAM-D) at post-treatment assessment, which measures severity of depression symptoms Total scores are displayed and represent summed scores on 17 individual items the scale, and scale range for total scores is 0 to 50.
  Higher scores indicate higher/worse levels of depression.
Time Frame: Post-Treatment assessment, occurring 12 weeks after the start of treatment (week 0)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Scores on a scale | 6.34 (6.00) | 11.84 (7.43)

6. Secondary Outcome: Hamilton Depression Scale (HAM-D) Total Score at 3-Month Follow-Up
Description: Hamilton Depression scale (HAM-D) at 3-month followup assessment, which measures severity of depression symptoms Total scores are displayed and represent summed scores on 17 individual items the scale, and scale range for total scores is 0 to 50.
  Higher scores indicate higher/worse levels of depression.
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Scores on a scale | 6.95 (7.39) | 11.45 (7.73)

7. Secondary Outcome: TLFB - Total Cigarettes Smoked Week Before Appointment (at Post-Treatment)
Description: Timeline Followback - Total number of cigarettes smoked the week before Post-Treatment visit
Time Frame: Week before Post-Treatment visit occurring at week 12, i.e. number of cigarettes smoked for the week prior to this week 12 visit
Measure: Mean (Standard Deviation); unit: Number of Cigarettes Smoked
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Number of Cigarettes Smoked | 14.31 (29.00) | 17.03 (28.15)

8. Secondary Outcome: TLFB - Cigarettes Smoked Week Before 3-Month Follow-up
Description: Timeline followback - Number of cigarettes smoked the week before 3-month follow-up visit
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: Number of Cigarettes Smoked
Arm/Group | Integrated Treatment | Varenicline
Number analyzed (Participants) | 72 | 70
Number of Cigarettes Smoked | 32.92 (45.64) | 25.85 (44.79)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire duration of data collection (2009-2015).
Description: Participants were assessed at each visit for adverse events (which typically occurred weekly).
Arm/Group | Integrated Treatment | Varenicline
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 6/72 | 4/70
Other Adverse Events (participants affected / at risk) | 64/72 | 58/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Treatment (N=72) | Varenicline (N=70)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Hospitalization secondary to drug or alcohol relapse (Surgical and medical procedures) | 1 (1) | 1 (1)
Respiratory issue (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) — Hospitalizations secondary to respiratory conditions (pneumonia, COPD, flu) for reasons unrelated to study procedures
Cocaine relapse with no hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Cocaine relapse with no hospitalization
Broken ankle + hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Broken ankle unrelated to study procedures that required hospitalization
Hospitalization (unrelated) (General disorders) | 0 (0) | 1 (1) — Reason for hospitalization unknown, but noted as unrelated to study procedures (general medical issue)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Integrated Treatment (N=72) | Varenicline (N=70)
Miscellaneous (General disorders) | 64 | 58 — Increased fatigue, increased/decreased appetite, dry mouth, diarrhea, etc

LIMITATIONS AND CAVEATS:
1. PPA verified by CO/cotinine was only assessed at two time-points (post-treatment, and follow-up)
2. medication adherence for varenicline was measured using pill count by the study nurse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes